CLINICAL TRIAL: NCT00071513
Title: Middle School to High School Transition Project
Brief Title: Middle School to High School Transition Project: Depression and Substance Abuse Prevention
Acronym: CAST-T/HSTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elizabeth McCauley, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21484-EG; R01MH061984 (NIH)
Record Dates: First submitted 2003-10-24; First posted 2003-10-28 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Depression; Substance-Related Disorders
Keywords: Adolescent; Substance Abuse; At-risk
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAST-T/HSTS (Experimental): The CAST-T/HSTS condition combined the Brief Intervention and 12 school based small group sessions which taught skills to enhance personal control (to manage depression, anger, stress), self-esteem, decision making and interpersonal communications. HSTS skills groups were held in the spring of 8th grade with 4 one-on-one booster sessions delivered to the students as 9th graders by HSTP leaders; parents also participated in 4 sessions. HSTS objectives are: 1) to increase the acquisition of coping skills competencies by teaching and practicing strategies taught; 2) to increase social support resources by building a supportive network; 3) to increase the youth's engagement in positive social activities; and 4) to motivate parents to increase their support via parent educational sessions.
  Interventions: Behavioral: CAST-T/HSTS
- Brief Intervention (Active Comparator): Brief Intervention: After each youth and parent completed baseline questionnaires the youth participated in a 1 on 1 standardized clinical follow-up with a trained clinician (blind to study condition) to review areas of concern, based on questionnaire responses including stressors at school, home, and with peers, level of support available and how to access support. The teen and clinician then planned a feedback call to parents, allowing teens to shape requests for support from parents as well as understand exactly what information would be shared with parents. Feedback call to parents reviewed concerns and made recommendations for services as needed. A similar procedure was followed after each assessment for all participants who indicated a risk of clinical depression or self-harm.
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: CAST-T/HSTS — Skills training small group.
  Arms: CAST-T/HSTS
Behavioral: Brief Intervention — Assessment of needs and referral to services as needed.
  Arms: Brief Intervention

SUMMARY:
This study will implement a school-based program to prevent depression, academic failure, and substance use in at-risk adolescents transitioning from middle school to high school.

DETAILED DESCRIPTION:
The transition from middle school to high school presents important challenges for adolescents. Programs that enhance personal efficacy and social support resources may prevent at-risk students from developing behaviors that can lead to substance use, academic failure, and depression. This study will implement a skills-based program called Coping and Support Training for the Transition (CAST-T) as a preventive intervention for at-risk students.

At-risk students in eighth grade will be randomly assigned to receive either CAST-T or school as usual. The CAST-T program will initially be delivered in twelve sessions over 6 weeks in the middle school setting. The program includes booster sessions, case management, structured home-based parent education, and support and skills training throughout the transition period. Participants will be assessed from the beginning of eighth grade to the end of ninth grade. Vulnerability to academic problems and depression will be assessed with school records and self-report scale scores.

ELIGIBILITY:
Inclusion Criteria:

* At-risk for substance abuse, academic failure, and depression
* Enrolled in eighth grade in Seattle Public Schools
* English-speaking

Exclusion Criteria:

* Score above the clinical cutoff on the Youth Self Report Aggressive subscale

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 497 (Actual)
Dates: Start 2003-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McCauley, PhD, Principal Investigator — University of Washington; Ann Vander Stoep, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Add data has been de-identified. De-identified data is available to share.

REFERENCES:
- [Background] Lyon AR, Ludwig KA, Stoep AV, Gudmundsen G, McCauley E. Patterns and Predictors of Mental Healthcare Utilization in Schools and other Service Sectors among Adolescents at Risk for Depression. School Ment Health. 2013 Aug 1;5(3):10.1007/s12310-012-9097-6. doi: 10.1007/s12310-012-9097-6. PMID 24223677
- [Background] Banh MK, Crane PK, Rhew I, Gudmundsen G, Stoep AV, Lyon A, McCauley E. Measurement equivalence across racial/ethnic groups of the mood and feelings questionnaire for childhood depression. J Abnorm Child Psychol. 2012 Apr;40(3):353-67. doi: 10.1007/s10802-011-9569-4. PMID 21996979
- [Background] Rhew IC, Simpson K, Tracy M, Lymp J, McCauley E, Tsuang D, Stoep AV. Criterion validity of the Short Mood and Feelings Questionnaire and one- and two-item depression screens in young adolescents. Child Adolesc Psychiatry Ment Health. 2010 Feb 9;4(1):8. doi: 10.1186/1753-2000-4-8. PMID 20181135
- [Background] Kuo E, Vander Stoep A, McCauley E, Kernic MA. Cost-effectiveness of a school-based emotional health screening program. J Sch Health. 2009 Jun;79(6):277-85. doi: 10.1111/j.1746-1561.2009.00410.x. PMID 19432868
- [Background] McCormick E, Thompson K, Stoep AV, McCauley E. The Case for School-Based Depression Screening: Evidence From Established Programs. Rep Emot Behav Disord Youth. 2009 Fall;9(4):91-96. PMID 26451134
- [Derived] Blossom JB, Adrian MC, Stoep AV, McCauley E. Mechanisms of Change in the Prevention of Depression: An Indicated School-Based Prevention Trial at the Transition to High School. J Am Acad Child Adolesc Psychiatry. 2020 Apr;59(4):541-551. doi: 10.1016/j.jaac.2019.05.031. Epub 2019 Jun 20. PMID 31228560
- [Derived] Makover H, Adrian M, Wilks C, Read K, Stoep AV, McCauley E. Indicated Prevention for Depression at the Transition to High School: Outcomes for Depression and Anxiety. Prev Sci. 2019 May;20(4):499-509. doi: 10.1007/s11121-019-01005-5. PMID 30852711
- See also: Project website — http://depts.washington.edu/pathways

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8th graders in 6 middle schools completed the screening battery; those with 15+ on the Moods and Feelings Questionnaire and below the clinical cutoff on the Youth Self Report, Aggressive subscale were eligible. 716 met criteria; 497 were randomized. 123 families or youth declined; the rest could not be contacted.
Pre-assignment Details: Participants recruited across 4 annual cohorts, included 241 youth randomized to HSTS and 256 to the Brief Intervention (BI). There were no significant differences between the 2 groups at baseline in terms of gender, race, and socioeconomic status (SES) as well as baseline comparisons of target variables (depression, hopelessness, anxiety, anger).
Groups:
- CAST-T/HSTS: HSTS condition combined the Brief Intervention and the HSTS protocol. HSTS introduced skills to enhance personal control (management of depression, anger and stress), self-esteem, decision making and interpersonal communications. Skills were taught in school based small groups to foster social support with outreach to teachers, peers, and parents. HSTS skills groups were held in the spring of 8th grade followed by four one-on-one booster sessions delivered to the students as 9th graders by HSTS leaders; parents participated in four educational sessions.
  HSTS objectives are: 1) to increase the acquisition of coping skills competencies by teaching and practicing strategies taught; 2) to increase social support resources by building a supportive network; 3) to increase the youth's engagement in positive social activities; and 4) to motivate parents to increase their support via parent educational sessions.
  CAST/HSTS Preventive Intervention: Brief Intervention
- Brief Intervention: Brief Intervention: After each youth and parent completed baseline questionnaires the youth participated in a 1 on 1 standardized clinical follow-up with a trained clinician (blind to study condition) to review areas of concern, based on questionnaire responses including stressors at school, home, and with peers, level of support available and how to access support. The teen and clinician then planned a feedback call to parents, allowing teens to shape requests for support from parents as well as understand exactly what information would be shared with parents. Feedback call to parents reviewed concerns and made recommendations for services as needed. A similar procedure was followed after each assessment for all participants who indicated a risk of clinical depression or self-harm.
  CAST/HSTS Preventive Intervention: Brief Intervention
Period: Intervention Component
Arm/Group | CAST-T/HSTS | Brief Intervention
Started | 241 | 256
Completed | 239 | 253
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Period: Follow-up Assessment
Arm/Group | CAST-T/HSTS | Brief Intervention
Started | 239 | 253
Completed | 233 | 247
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- CAST-T/HSTS: HSTS condition combined the Brief Intervention and the HSTS protocol. HSTS introduced skills to enhance personal control (management of depression, anger and stress), self-esteem, decision making and interpersonal communications. Skills were taught in school based small groups to foster social support with outreach to teachers, peers, and parents. HSTS skills groups were held in the spring of 8th grade followed by four one-on-one booster sessions delivered to the students as 9th graders by HSTP leaders; parents participated in four educational sessions.
  HSTS objectives are: 1) to increase the acquisition of coping skills competencies by teaching and practicing strategies taught; 2) to increase social support resources by building a supportive network; 3) to increase the youth's engagement in positive social activities; and 4) to motivate parents to increase their support via parent educational sessions.
  CAST/HSTS Preventive Intervention: Brief Intervention
- Total: Total of all reporting groups
Arm/Group | CAST-T/HSTS | Brief Intervention | Total
Number analyzed (Participants) | 241 | 256 | 497
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 241 | 256 | 497
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (0.83) | 13.65 (0.67) | 13.57 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 165 | 314
  Male | 92 | 91 | 183
Region of Enrollment [Number; unit: participants]
  United States | 241 | 256 | 497

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Moods and Feelings Questionnaire (SMFQ)
Description: The Short Moods and Feelings Questionnaire is a 13 item measure of level of self reported depressive symptoms. Each item in scored on a 3-point Likert scale as follows: "True" (0), "Sometimes" (1), and "Not True" (2) rated within the timeframe of the previous two weeks. A total score is obtained; scores can range from 0 to 26. Total scores of 12 or higher may signify that a child/adolescent is suffering from depression. Higher scores on this scale suggest a worse outcome or greater endorsement of depressive symptoms. Change is measured based on two time points baseline to the 18 months follow-up assessment.
Time Frame: Baseline to 18 months
Population: The main study hypothesis was that at-risk middle school students randomly assigned to participate in the CAST-T/HSTS versus the Brief Intervention would demonstrate a greater reduction in self-reported depressive symptoms after the 8th grade intervention as well as lower rate of increase in depressive symptoms at the 18 mos. follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAST-T/HSTS | Brief Intervention
Number analyzed (Participants) | 233 | 247
units on a scale | 2.19 (6.18) | 1.21 (6.40)
Statistical Analysis 1: Comparison: CAST-T/HSTS vs Brief Intervention; Mean changes in Short Moods and Feelings measure of depression was the unit of analysis; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: CAST-T/HSTS vs Brief Intervention; A secondary hypothesis of the study was that attachment to school and/or perceptions of school supportiveness would mediate the effect of the HSTS intervention on depressive symptoms; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: School Attachment
Description: School attachment measure consisted of 4 items. Item responses range from 0 (unsatisfied, rarely attended, not involved, etc.) to 6 (highly satisfied, regularly attended, very involved, etc). Scores could range from 0 to 36 with higher scores indicating more positive school attachment. Item were:
  My overall satisfaction with classes was… Overall, how safe did school feel last semester… Overall, how friendly did school feel… How involved were you in school activities…
Time Frame: 18 months
Population: T-test differences for HSTS versus Brief Intervention on the School Attachment scale.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | CAST-T/HSTS | Brief Intervention
Number analyzed (Participants) | 233 | 247
units of a scale | 4.53 (1.21) | 3.95 (1.31)

ADVERSE EVENTS:
Time Frame: 18 months, from initial screening which began in January of the 8th grade year to final follow-up assessments which were conducted in spring of the ith grade year (April to June) approximately 18 months later.
Description: At baseline each youth was interviewed by a trained clinician with a feedback call to parents. Thereafter, at each assessment, any student with responses indicating risk of clinical depression or self-harm was immediately assessed by a clinical specialist who worked with parents and the school counselors to develop an intervention/support plan.
Arm/Group | CAST-T/HSTS | Brief Intervention
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/256
Other Adverse Events (participants affected / at risk) | 0/241 | 0/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAST-T/HSTS (N=241) | Brief Intervention (N=256)
Severe depression and/or suicidal risk requiring immediate intervention (Psychiatric disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A significant limitation of this trial was the brief nature of the comparison condition, the Brief Intervention group; findings might reflect "dose" rather than content of the CAST-T/HSTS intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes